CLINICAL TRIAL: NCT00313521
Title: Continuous Infusion Thiotepa in High Grade Astrocytic Tumors of Childhood and Adolescence A UKCCSG Phase II Study Involving the Brain Tumour and New Agent Groups
Brief Title: Thiotepa and Radiation Therapy in Treating Young Patients With Newly Diagnosed Malignant Brain Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000454503; CCLG-9405; EU-20575; CCLG-CNS-1995-01
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2006-12

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: untreated childhood cerebellar astrocytoma; childhood high-grade cerebral astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma | interventions — Thiotepa; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Drug: thiotepa
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as thiotepa, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving chemotherapy and radiation therapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well thiotepa works together with radiation therapy in treating young patients with newly diagnosed malignant brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine tumor response to adjuvant thiotepa followed by radiotherapy in pediatric patients with newly diagnosed malignant astrocytic tumors.

Secondary

* Determine the acute and chronic toxicity of thiotepa in these patients.
* Determine the variability in thiotepa metabolism by measuring plasma and cerebrospinal fluid pharmacokinetics of thiotepa and tepa in these patients.
* Develop a phase II study framework model, to determine the chemosensitivity to new, single-agent regimens in the treatment of high-grade (malignant) astrocytic tumors, including anaplastic astrocytoma, glioblastoma, giant cell glioblastoma, and gliosarcoma.
* Determine the incidence of distant neuraxial metastases in patients at the time of relapse.
* Determine the 1-year disease-free survival rate in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified by age (3-15 vs 16-20 years of age).

* Chemotherapy: Patients receive thiotepa IV continuously over 168 hours on days 1-7. Treatment repeats every 28 days for up to 2 courses. Patients then proceed to radiotherapy after blood counts recover.
* Radiotherapy: Patients undergo external-beam radiotherapy once daily, 5 days a week, for approximately 6 weeks.
* Post-radiation chemotherapy: Patients with complete, partial, or objective response, or stable disease after 2 courses of thiotepa may receive thiotepa alone for up to 8 more courses at the discretion of the treating physician.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following high-grade (malignant) astrocytic tumors:

  * Anaplastic astrocytoma
  * Glioblastoma
  * Giant cell glioblastoma
  * Gliosarcoma
* Any anatomical site except brain stem
* Newly diagnosed disease
* Has undergone tumor biopsy or surgical resection within the past 2 weeks

  * Patients with post-operative residual disease (grade III or IV) are eligible

    * Post-operative imaging of tumor within 72 hours of surgery
  * Patients with no imageable post-operative disease are not eligible
* No neurological deterioration within 3 days of study treatment

  * Increasing requirement for steroids to control symptoms of intracranial pressure is considered evidence of neurological deterioration

PATIENT CHARACTERISTICS:

* Lansky play score 40-100%
* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3
* Creatinine ≥ 1.5 times upper limit of normal

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy or radiotherapy

Ages: 3 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 1995-06; Primary Completion 1997-11 (Estimated)

PRIMARY OUTCOMES:
Degree of surgical resection by surgical and radiological assessments

SECONDARY OUTCOMES:
Tumor response to chemotherapy by imaging

CONTACTS AND LOCATIONS:
Overall Officials: David A. Walker, Study Chair — Queen's Medical Center